CLINICAL TRIAL: NCT04973098
Title: An Open-Label, Dose Escalation/Dose Exploration, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single/Multiple Infusion of CT0181 Injection in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Phase I Clinical Trial of CT0181 Cells in the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0181-CG1202
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Carcinoma; Hepatocellular Neoplasms
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5 dose levels each with or without lymphocyte clearance were tentatively determined. (Experimental): CT0181 Cells were transfused after lymphocyte clearance with fludarabine and cyclophosphamide or without lymphocyte clearance.
  Interventions: Biological: CT0181 Cells

INTERVENTIONS:
Biological: CT0181 Cells — 5 dose levels each with or without lymphocyte clearance were tentatively determined.
  Other Names: CT0181 humanized anti GPC3 autogenous T Cell injection

SUMMARY:
A Phase I Clinical Study of CT0181 cells in Patients with Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
Primary objectives:

Evaluate the safety and tolerance of CT0181 cells in patients with advanced hepatocellular carcinoma within 28 days after the first infusion

Secondary objectives:

Evaluate the metabolic kinetics of CT0181 cells ; Evaluate overall safety and tolerability ; Evaluate the initial efficacy of CT0181 cell infusion in the treatment of advanced hepatocellular carcinoma with positive Glypican-3（GPC3 ）expression.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, either sex；
2. Patients with clinically or pathologically confirmed hepatocellular carcinoma were treated with surgery or local treatment It is not suitable for surgery or local radical treatment;
3. Progression or intolerance after at least one previous systemic treatment, or due to specific reasons unable to receive systemic treatment.
4. According to Barcelona Clinic Liver Cancer（BCLC）, the patients are classified into Grade C or Grade B unsuitable for local treatment/progressive disease after local treatment;
5. In tumor tissue samples GPC3 is detected positive by immunohistochemistry (IHC);
6. According to Response Evaluation Criteria in SolidTumors（RECIST1.1）,patients have at least one evaluable target lesion;
7. Expected survival is > 12 weeks;
8. Cirrhosis status Child-Pugh score: ≤7
9. Eastern Cooperative Oncology Group Performance Status score: 0 to 1 point;
10. If the patient is HBsAg positive or HBcAb positive, DNA of the hepatitis B virus should be <2000 IU/ml. HBsAg positive patients must receive antiviral treatment ;
11. Acceptable routine blood test showing no contraindication to the lymphodepletion pretreatment and adequate liver, renal, cardiovascular, respiratory function;
12. Have venous accesses for apheresis;
13. Subjects of childbearing age must undergo a serum pregnancy test . In addition, they should be willing to use a reliable method of contraception during the trial (within 52 weeks after cell infusion); male subjects whose spouses are women of childbearing age should undergo sterilization surgery or agree to use a reliable method of contraception during the trial; Understand and sign informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. Hepatitis virus C antibodies ,Human Immunodeficiency Virus（HIV） antibodies or Syphilis Serological tests are positive;
3. Any uncontrol active infection, including but not limited to active tuberculosis;
4. Have clinically significant thyroid dysfunction except the stable control after treatment;
5. Previous or present hepatic encephalopathy;
6. Current clinically significant ascites;
7. Imaging results:≥50% of the liver is replaced by tumor or portal vein main tumor thrombus, or metastases to the central nervous system, or tumor thrombus invasion of mesenteric vein / inferior vena cava;
8. Subjects have known active autoimmune diseases
9. The side effects caused by the previous treatment of the subjects did not return to Common Terminology Criteria for Adverse Events（CTCAE） ≤1; except hair loss and other tolerable events determined by investigator;
10. Patients who had received systemic steroids or other immunosuppressive agents within 7 days before apheresis, except inhaled steroids;
11. History of severe allergy ;
12. Has signs of central nervous system disease or an abnormal neurological examination with clinical significance;
13. Subjects with unstable or active ulcers, gastrointestinal bleeding, or pump inhibitor intolerance;
14. Patients with a history of organ transplantation or waiting for organ transplantation;
15. Previously received Programmed cell Death-1/Programmed cell Death-Ligand 1 monoclonal antibody therapy within 4 weeks or local treatment and systemic chemiotherapy within 2 weeks or immunotheray and molecular targeted drugs within 1 week before apheresis;
16. Previously received GPC3 targeted therapy;
17. Major surgery or significant trauma occurred within 4 weeks before apheresis, or it is expected that major surgery needs to be performed during the trial;
18. Patients who had incurable malignant tumors in the past 5 years or at the same time, except cervical cancer in situ and basal cell carcinoma of skin;
19. Other serious diseases that may restrict the subjects from participating in the trial ；
20. The researcher assessed that the subjects were unable or unwilling to comply with the requirements of the trial protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
1.Dose-Limiting Toxicity（DLT） | 28days
  Safety
Maximal Tolerable Dose（MTD） | 28days
  tolerability evaluation
Treatment Emergent Adverse Event（TEAE） | 28days
  Incidence rate
Adverse Event of Special Interest | 28 days
  Incidence rate

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No